CLINICAL TRIAL: NCT04910438
Title: Prevalence and Longitudinal Follow-up Over 2 Years of Anal Lesions, HPV Infection and Associated Sexually Transmitted Infections Among Men Who Have Sex With Men (MSM) in Lomé, Togo
Brief Title: Prevalence and Longitudinal Follow-up of Anal Lesions, HPV Infection and Associated Sexually Transmitted Infections Among Men Who Have Sex With Men in Togo.
Acronym: DepIST-H
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Université de Lomé, Département de Santé Publique, Lomé, Togo (Unknown); Bichat Hospital (Other); Espoir Vie-Togo - ONG (Other); Centre Africain de Recherche en Epidémiologie et en Santé Publique, Lomé, Togo (Unknown); Programme PAC-CI, Site ANRS-MIE de Côte d'Ivoire (Other); Laboratoire de Biologie Moléculaire et d'Immunologie, Lomé, Togo (Unknown); Saint-Louis Hospital, Paris, France (Other); University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: ANRS 12400 DepIST-H
Record Dates: First submitted 2020-01-22; First posted 2021-06-02 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Papillomavirus Infections; HIV Infections
Keywords: HPV; HIV; MSM; Togo
MeSH Terms: conditions — Papillomavirus Infections; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, Blood Anal smear pharyngeal and oral specimens urethral specimens Swab of herpes vesicles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: STIs screening and care — * Screening for anal dysplasia, HPV infection, HIV infection and several STIs (Neisseria gonorrhoeae, Chlamydia trachomatis, Mycoplasma genitalium, Trichomonas vaginalis, HSV-2 and HBV).
  * Offering comprehensive care including prevention strategies adapted to the various STIs mentioned above and their complications, particularly the progression to anal cancer for HPV infections in MSM.

SUMMARY:
The DepIST-H study, funded by the French AIDS and Hepatitis Research Agency (ANRS), is to estimate prevalence (the number of cases over a given period of time) and incidence (the number of new cases over a given period of time) of anal lesions (condylomas, dysplasia, cancers) by HIV status among MSM in Lomé, Togo

DETAILED DESCRIPTION:
Title: Prevalence and longitudinal follow-up over 2 years of anal lesions, HPV infection and associated sexually transmitted infections among men who have sex with men (MSM) in Lomé, Togo (ANRS12400 DepIST-H)

Main objective: To estimate the prevalence and incidence of anal lesions (condyloma, dysplasia and anal cancers) according to HIV status among MSM in Lomé, Togo

Specific objectives :

To estimate the prevalence of HPV infection at baseline (M0) at anal and oropharyngeal sites To describe the persistence of HPV infection at Year 1 and 2 at the anal and oropharyngeal sites To describe the recurrence of anal lesions at Year 1 and 2 To estimate prevalence and incidence of associated STIs (Neisseria gonorrhoeae, Chlamydia trachomatis, Herpes simplex Virus type 2, Mycoplasma genitalium, Trichomonas vaginalis) HBV, HCV and syphilis

Methods :

This study is a prospective cohort with a 2-year follow-up of 200 MSM in Lomé (100 HIV- and 100 HIV+). Three data collection systems are integrated into the cohort: (i) clinical data, (ii) socio-behavioural questionnaires, and (iii) biological data.

Sample size: 200 participants (100 HIV+ and 100 HIV-)

Interventions :

Screening for anal dysplasia, HPV infection, HIV infection and several STIs (Neisseria gonorrhoeae, Chlamydia trachomatis, Mycoplasma genitalium, Trichomonas vaginalis, HSV-2 and HBV).

Offering comprehensive care including prevention strategies adapted to the various STIs mentioned above and their complications, particularly the progression to anal cancer for HPV infections in MSM.

Statistical analysis methods :

Use of mixed approaches. For quantitative indicators, descriptive analysis techniques, bivariate analysis (Student t test or Wilcoxon test for quantitative variables, Chi² or Fisher test for categorical variables) and multivariate analysis (logistic regression).

To estimate the incidence if the STIs, Kaplan-Meier curves, Cox models analyses will be conducted.

As the cohort is open and non-randomized, preliminary analyses will be conducted during the collection.

ELIGIBILITY:
Inclusion Criteria:

* Being a male aged 18 or over
* Self-reporting as being a MSM
* Wishing to be part of a regular clinical follow-up
* Agreeing to participate in the study and signing the informed consent form
* Live in Lomé
* Having had anal intercourse within the past six months prior to inclusion visit
* Regardless of HIV status (infected or not)
* Whether or not the participant has already taken antiretrovirals

Exclusion Criteria:

* Participation in another biomedical and/or behavioural study on HIV, viral hepatitis or sexually transmitted infections (CohMSM ANRS 12324-EF cohort of Lomé)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male who have sex with men living with HIV or not
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence at inclusion of anal lesions | at Day 0
  According to HIV status among MSM in Lomé, Togo

SECONDARY OUTCOMES:
Prevalence of anal lesions at baseline | at Day 0
  According to HIV status among MSM in Lomé, Togo
Incidence of anal lesions | at 12 month and 24 month
  According to HIV status among MSM in Lomé, Togo
Describe the number of worsening events of anal cytological lesions | at 12 month and 24 month
  According to HIV status among MSM in Lomé, Togo
Describe the proportion of recurrence of anal lesions | at 12 month and 24 month
  According to HIV status among MSM who received available treatment, in Lomé, Togo
Prevalence of HPV infections | at Day 0
Incidence of HPV infection | at 12 month and 24 month
Describe the proportion of persistent HPV infections | at 12 month and 24 month
Describe the proportion of clearance of HPV infections | at 12 month and 24 month
  in the same individual, on anal and oral specimens, based on HIV status.

OTHER OUTCOMES:
Prevalence of others STIs : N. gonorrhoeae, C. trachomatis, M. genitalium, T. vaginalis, Herpès Simplex Virus type 2 (HSV-2), syphilis, hepatitis B and hepatitis C | At Day 0, at 12 month and 24 month
  According to HIV status
Incidence of others STIs : Neisseria gonorrhoeae, Chlamydia trachomatis, Mycoplasma genitalium, Trichomonas vaginalis and Herpès Simplex Virus type 2 (HSV-2), syphilis, hepatitis B and hepatitis C | At Day 0, at 12 month and 24 month
  According to HIV status
Determination of different Chlamydia trachomatis strains | At Day 0
Determination of antibiotic resistance profiles for Neisseria gonorrhoeae, Mycoplasma genitalium and Chlamydia trachomatis | At Day 0
  According to HIV status
Incidence of HIV | at 12 month and 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Charpentier, Principal Investigator — Hôpital Bichat Claude Bernard, Paris, France; Didier Ekouevi, Principal Investigator — Lomé University, Togo
Locations (1):
- ONG, Espoir Vie Togo, Lomé, Togo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferre VM, Sadio AJ, Gbeasor-Komlanvi FA, Bucau M, Salou M, Bercot B, Bebear C, Abramowitz L, Zaidi M, Amenyah-Ehlan AP, Mensah E, Braille A, Couvelard A, Dagnra AC, Ghosn J, Descamps D, Charpentier C, Ekouevi DK. High prevalence of bacterial STI, anal HPV, cytological abnormalities and anal lesions among MSM in Togo, 2021: a baseline analysis of the ANRS I MIE 12,400/DepIST-H cohort. BMC Infect Dis. 2025 Sep 26;25(1):1156. doi: 10.1186/s12879-025-11338-y. PMID 41013315